CLINICAL TRIAL: NCT02848066
Title: Open, Parallel, Single-Site Study to Evaluate Sensitivity and Specificity of Newly Defined Diagnosed-biomarker for Gastric Cancer Pts and Cancer-free Healthy Volunteers
Brief Title: Glycans Bound to Serum Haptoglobin: a Novel Gastric Cancer Tumor Biomarker
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-07-146
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastric Cancer patients: This arm is composed of the gastric cancer patients. It is perfomed a blood sampling to them after the research registration.
  Interventions: Procedure: Blood sample(10cc) collection
- Cancer-free healthy volunteers: This arm is composed of the cancer-free healthy volunteers. It is perfomed a blood sampling to them after the research registration.
  Interventions: Procedure: Blood sample(10cc) collection

INTERVENTIONS:
Procedure: Blood sample(10cc) collection — In both groups, serum haptoglobins to be collected and analyzed

SUMMARY:
The purpose of this study is to evaluate sensitivity and specificity of newly defined tumor biomarker with gastric cancer pts and cancer-free healthy volunteers.

DETAILED DESCRIPTION:
Measurements of specific glycosylation changes in serum haptoglobin.

ELIGIBILITY:
Arm1 (Gastric cancer patient)

1. Inclusion Criteria:

   * Male or female over 19 years
   * Patients with histologically Gastric Cancer (included Gastroesphageal junction)
   * Primary gastric cancer or/and metastatic gastric cancer.
   * Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
2. Exclusion Criteria:

   * Prior or present history of malignancies other than gastric cancer
   * Any condition that confounds the ability to interpret data from the study under the investigational confirmed.

Arm2 (Cancer-free healthy volunteers)

1. Inclusion Criteria:

   * Male or female over 19 years
   * Cancer-free status.
   * Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
2. Exclusion Criteria:

   * Prior or present history of malignancies (included gastric cancer)
   * Any condition that confounds the ability to interpret data from the study under the investigational confirmed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Arm1- Gastric cancer patient: 150 subjects Arm2- Cancer-free healthy volunteers : 203
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
AUC(Area Under the Curve) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Relative abundance of glycosylations | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etzioni R, Urban N, Ramsey S, McIntosh M, Schwartz S, Reid B, Radich J, Anderson G, Hartwell L. The case for early detection. Nat Rev Cancer. 2003 Apr;3(4):243-52. doi: 10.1038/nrc1041. PMID 12671663
- [Background] Paik YK, Kim H, Lee EY, Kwon MS, Cho SY. Overview and introduction to clinical proteomics. Methods Mol Biol. 2008;428:1-31. doi: 10.1007/978-1-59745-117-8_1. PMID 18287765
- [Background] Asazawa H, Kamada Y, Takeda Y, Takamatsu S, Shinzaki S, Kim Y, Nezu R, Kuzushita N, Mita E, Kato M, Miyoshi E. Serum fucosylated haptoglobin in chronic liver diseases as a potential biomarker of hepatocellular carcinoma development. Clin Chem Lab Med. 2015 Jan;53(1):95-102. doi: 10.1515/cclm-2014-0427. PMID 25060348
- [Background] Hoagland LF 4th, Campa MJ, Gottlin EB, Herndon JE 2nd, Patz EF Jr. Haptoglobin and posttranslational glycan-modified derivatives as serum biomarkers for the diagnosis of nonsmall cell lung cancer. Cancer. 2007 Nov 15;110(10):2260-8. doi: 10.1002/cncr.23049. PMID 17918261
- [Background] Thompson S, Cantwell BM, Matta KL, Turner GA. Parallel changes in the blood levels of abnormally-fucosylated haptoglobin and alpha 1,3 fucosyltransferase in relationship to tumour burden: more evidence for a disturbance of fucose metabolism in cancer. Cancer Lett. 1992 Aug 14;65(2):115-21. doi: 10.1016/0304-3835(92)90154-n. PMID 1511415
- [Background] Park SY, Lee SH, Kawasaki N, Itoh S, Kang K, Hee Ryu S, Hashii N, Kim JM, Kim JY, Hoe Kim J. alpha1-3/4 fucosylation at Asn 241 of beta-haptoglobin is a novel marker for colon cancer: a combinatorial approach for development of glycan biomarkers. Int J Cancer. 2012 May 15;130(10):2366-76. doi: 10.1002/ijc.26288. Epub 2011 Sep 22. PMID 21780104
- [Background] Dennis JW, Granovsky M, Warren CE. Glycoprotein glycosylation and cancer progression. Biochim Biophys Acta. 1999 Dec 6;1473(1):21-34. doi: 10.1016/s0304-4165(99)00167-1. PMID 10580127